CLINICAL TRIAL: NCT00129558
Title: A Phase I/II Study of PT-523 in Patients With Refractory Leukemia
Brief Title: A Study to Evaluate PT-523 in Patients With Refractory Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: HBS103
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — N(alpha)-(4-amino-4-deoxypteroyl)-N(delta)-hemiphthaloyl-L-ornithine; Injections

INTERVENTIONS:
Drug: PT-523 for Injection

SUMMARY:
This Phase I/II, multi-centered, non-randomized, trial is designed to determine a safe dose of PT-523 for subjects, and to make preliminary evaluations on the activity of PT-523 as therapy in subjects with refractory leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed/refractory leukemias including acute non-lymphocytic leukemia (AML), acute lymphocytic leukemia (ALL), chronic lymphocytic leukemia (CLL), and chronic myelogenous leukemia in blastic phase (CML-BP) for which no standard therapies are anticipated to result in a durable remission; or poor-risk myelodysplasia (MDS) patients to include refractory anemia with excess blasts (RAEB) or excess blasts in transformation (RAEBT) and chronic myelomonocytic leukemia (CMML) who are either relapsed/refractory or who refuse/are not eligible for frontline therapy.
* Only patients with refractory ALL or CML in lymphoid blastic phase are eligible for phase II.
* ECOG performance status 0 - 2.
* Adequate organ function and bone marrow reserve.
* At least 4 weeks must have elapsed from the time of major surgery.
* Use of appropriate contraceptive method.
* Signed patient informed consent.

Exclusion Criteria:

* Known human immunodeficiency virus (HIV).
* Active heart disease including myocardial infarction within previous 3 months, symptomatic coronary artery disease, arrhythmias not controlled by medication, or uncontrolled congestive heart failure.
* Patients receiving any other standard or investigational treatment for their leukemia other than corticosteriods, hydroxyurea, and 6-mercaptopurine.
* Any medical condition which, in the opinion of the investigator, places the patient at an unacceptably high risk for toxicities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - USC, Kennth Norris Jr. Comprehensive Cancer Center, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine Comprehensive Cancer Center, Winston-Salem, North Carolina
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: Hana Biosciences, Inc. is a South San Francisco, CA-based biopharmaceutical company that acquires, develops, and commercializes innovative products to advance cancer care. — http://www.hanabiosciences.com